CLINICAL TRIAL: NCT04740697
Title: Pilot Study to Evaluate the Impact of the Use of Alternative and Complementary Therapies on Therapeutic Adherence in Patients Treated With taMoxifen for Early Stage Breast Cancer
Brief Title: Study to Evaluate the Impact of the Use of Alternative and Complementary Therapies on Therapeutic Adherence in Patients Treated With taMoxifen for Early Stage Breast Cancer
Acronym: EUTACAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20 SEIN 13
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Tamoxifen; Alternative and complementary therapies; Treatment adherence; Turmeric
MeSH Terms: conditions — Breast Neoplasms; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with localized breast cancer. (Other)
  Interventions: Other: Treatment requiring adjuvant Hormonal Therapy (HT) with tamoxifen.

INTERVENTIONS:
Other: Treatment requiring adjuvant Hormonal Therapy (HT) with tamoxifen. — Each included patient will be referred to the health care staff for a blood sample:
  * for the determination of the residual plasma concentration of tamoxifen and its active metabolites,
  * for the constitution of a biobank.
  Patients will then complete a questionnaire to collect information on tamoxifen intake and adherence (via the GIRERD questionnaire), as well as possible Alternative and Complementary Therapeutics (ACT) intake (reason for use, type of ACT, ...).

SUMMARY:
This is a pilot, prospective, interventional, monocentric study designed to evaluate, in a real-life situation, adherence to tamoxifen treatment as a function of the taking of alternative and complementary therapies in patients with localized hormone-dependent breast cancer.

200 patients will be included in the study.

Each patient will be followed for one day.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at entry into the study.
2. Patient treated for hormone-dependent localized breast cancer requiring adjuvant Hormonal Therapy (HT) with tamoxifen.
3. Patients treated with tamoxifen for a maximum of 1 to 3 years.
4. Patient affiliated with a Social Security system in France.
5. Patients who signed informed consent prior to inclusion in the study and prior to any specific study procedures.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Any psychological, family, geographical or sociological condition that does not allow the medical follow-up and/or the procedures foreseen in the study protocol to be respected.
3. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who adhere to tamoxifen treatment. | 18 months after the start of the research
  This outcome will be assessed by the completion of the GIRERD questionnaire by the patient.

SECONDARY OUTCOMES:
Rate of patients taking ACT. | 18 months after the start of the research
Rate of patients consuming turmeric-based dietary supplements. | 18 months after the start of the research
Plasma concentration of tamoxifen in patients. | 18 months after the start of the research

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France